CLINICAL TRIAL: NCT03631641
Title: A Phase II Study of PD-1 Inhibition for the Prevention of Colon Adenomas in Patients With Lynch Syndrome and a History of Partial Colectomy
Brief Title: Nivolumab in Preventing Colon Adenomas in Participants With Lynch Syndrome and a History of Partial Colectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: John Hays (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, John Hays, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSU-17198; NCI-2018-01491 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Colon Adenoma; Colon Carcinoma; Lynch Syndrome; MLH1 Gene Mutation; MSH2 Gene Mutation
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Participants receive nivolumab intravenously IV over 60 minutes on day 1. Treatment repeats every 3 months for a total of 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab works in preventing colon adenomas in participants with Lynch syndrome and a history of surgery to remove part of the colon. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if maintenance therapy with nivolumab can decrease the incidence of colon adenomas in a population of patients with genetic predisposition to colorectal cancer and a history of hemicolectomy due to colon cancer or advanced colon adenoma.

SECONDARY OBJECTIVES:

I. To assess the safety of nivolumab maintenance therapy in this population. II. To obtain preliminary data on the short-term incidence of advanced colon adenomas (measuring greater than 10 mm or with high-grade dysplasia) and colon and non-colonic cancers in Lynch patients treated with maintenance nivolumab.

EXPLORATORY OBJECTIVES:

I. To determine biomarkers of immunologic activity associated with biologic activity of nivolumab in this population.

OUTLINE:

Participants receive nivolumab intravenously (IV) over 60 minutes on day 1. Treatment repeats every 3 months for a total of 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 3 months, every 6 months for 1 year, then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a diagnosis of Lynch syndrome confirmed by the identification of a germline mutation in MLH1 or MSH2.
* Patient must have a history of colon cancer or advanced colon adenoma requiring hemicolectomy with at least 60 cm of colon remaining without evidence of disease.
* Be willing and able to provide written informed consent/assent for the trial.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Absolute neutrophil count (ANC) >= 1,500 /mcL within 10 days of treatment initiation.
* Platelets >= 100,000 / mcL within 10 days of treatment initiation.
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency within 10 days of treatment initiation.
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN within 10 days of treatment initiation.
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN within 10 days of treatment initiation.
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases within 10 days of treatment initiation.
* Albumin >= 2.5 mg/dL within 10 days of treatment initiation.
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants within 10 days of treatment initiation.
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants within 10 days of treatment initiation.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug.
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with nivolumab plus 5 half-lives of nivolumab (19 weeks) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks post-treatment completion.
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with nivolumab plus 5 half-lives of the study drug (19 weeks) plus 90 days (duration of sperm turnover) for a total of 31 weeks post-treatment completion.
* Hemicolectomy and adjuvant chemotherapy (if given) must be completed at least one year prior to study entry.
* All subjects must take at least 81 mg of aspirin per day. Daily doses up to 650 mg of aspirin per day will be accepted.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Individuals who are receiving systemic steroid therapy at a stable dose less than or equal to 10 mg of prednisone per day or its equivalent will be permitted to participate.
* Has a known history of active TB (Bacillus tuberculosis).
* Hypersensitivity to nivolumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had hemicolectomy, prior chemotherapy, targeted small molecule therapy, or radiation therapy within one year prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with =< grade 2 neuropathy and/or alopecia are an exception to this criterion and may qualify for the study.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids exceeding 10 mg prednisone per day or its equivalent, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of, active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Have a known history of a bleeding disorder or gastrointestinal ulceration that would preclude the use of a daily 81 mg aspirin.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or is expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* Subjects with germline MSH6, PMS2, or EPCAM mutations will be excluded from participation.
* Prisoners or individuals who are compulsorily detained will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hays, MD, Ph.D, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Adenomas
Description: The associated confidence intervals will be reported and used to determine if the incidence rate is significantly different from that reported among Lynch patients not receiving nivolumab, 0.33.
Time Frame: At 3 years
Population: Data was not obtained and analyzed due to early study termination
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

2. Primary Outcome: Incidence Rate of High-risk Adenomas
Description: The associated confidence interval will be reported and used to determine if the incidence rate is significantly different from 0.22, the reported incidence of high-risk adenomas among Lynch syndrome patients not receiving nivolumab.
Time Frame: At 3 years
Population: Data was not obtained and analyzed due to early study termination
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

3. Primary Outcome: Incidence Rate of Colon Cancers
Description: The incidence rates of colon cancers in Lynch patients treated with nivolumab will be estimated with corresponding confidence intervals.
Time Frame: At 3 years
Population: Data was not obtained and analyzed due to early study termination
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

4. Primary Outcome: Incidence Rate of Non-colonic Cancers
Description: The incidence rates of non-colonic cancers in Lynch patients treated with nivolumab will be estimated with corresponding confidence intervals.
Time Frame: At 3 years
Population: Data was not obtained and analyzed due to early study termination
Arm/Group | Treatment (Nivolumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse experiences will be graded and recorded throughout the study and during the follow-up period according, an average of 2 years.
Arm/Group | Treatment (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab) (N=3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Bilateral skin lesions- arms and legs- 1 lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
decreased eGFR (Renal and urinary disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear Pain (left ear) radiating with headmovment (Ear and labyrinth disorders) | 1 (1)
eczema- bilateral hands (Skin and subcutaneous tissue disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
fever (General disorders) | 1 (1)
Glucose Intolerance (Metabolism and nutrition disorders) | 2 (2)
heart palpitations (Cardiac disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Localized Edema-Left Calf (General disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
menorrhagia (Reproductive system and breast disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
neuropathy bilateral fingers (Nervous system disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (2)
Seborrheic Keratosis (1 forearm lesion) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Lesions (Skin and subcutaneous tissue disorders) | 2 (2)
squamous cell ca-5 lesions-bilateral arms and legs (Skin and subcutaneous tissue disorders) | 1 (1)
transient thyroiditis (Endocrine disorders) | 1 (1)
TSH decreased (Endocrine disorders) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1)
weight loss (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial stopped early due to withdrawal of pharmaceutical sponsor support

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03631641/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03631641/ICF_002.pdf